CLINICAL TRIAL: NCT06165887
Title: The Relationship Between Moderate-to-severe Psoriasis and Sleep Disturbance: a Prospective Cohort Study
Brief Title: The Relationship Between Moderate-to-severe Psoriasis and Sleep Disturbance
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20231008
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Moderate-to-severe Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate-to-severe Psoriasis patients: Participants will fill out questionnaires to assess sleep status and the severity of psoriasis.
  Interventions: Other: No intervention
- Healthy people: Participants will fill out questionnaires to assess sleep status
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study, no intervention will be implemented.
  Groups: Moderate-to-severe Psoriasis patients
Other: No intervention — This is an observational study, no intervention will be implemented.
  Groups: Healthy people

SUMMARY:
Psoriasis is a common chronic and systemic immune-mediated disease, induced by a combination of genetic and environmental effects. The increasingly worrying question is the negative impact on patients' sleep, which has become an important comorbidity of psoriasis. To investigate the causal relationship between psoriasis and sleep status, a prospective cohort study will be conducted by separating moderate-to-severe psoriasis patients and healthy individuals into distinct cohorts in order to observe their sleep status.

DETAILED DESCRIPTION:
Target follow-up duration for the study is 24 weeks, during which participants will undergo a sleep monitoring session every 8 weeks. The sleep monitoring data collected includes time to fall asleep, time to bed, sleep perception, and the Pittsburgh Sleep Quality Index (PSQI). The Dermatology Quality of Life Index (DLQI), the Psoriasis Area and Severity Index (PASI), and the Visual Analog Scale (VAS) will simultaneously be used to assess the severity of the disease in the cohort of patients with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. In line with the diagnostic criteria of psoriasis
2. PASI>10 or BSA>10%
3. Understand and agree to participate in this study and sign the informed consent.

Exclusion Criteria:

1. Those with serious mental diseases, such as depression, anxiety, etc;
2. PSQI>5 points;
3. Long term use of sedative and hypnotic drugs;
4. Patients with diabetes mellitus or severe heart, liver and kidney disease;
5. Those diagnosed with sleep disorders, such as apnea syndrome, periodic limb movement disorder, restless legs syndrome, narcolepsy, etc;
6. There are serious cardiovascular and cerebrovascular diseases, respiratory system diseases, and immune system diseases;
7. Pregnant women during pregnancy, lactation, or planned trials;
8. Those who have participated in other clinical studies or are participating in other clinical trials within 3 months;
9. Unable to cooperate with the study for any reason, such as the following situation: language understanding, unable to complete the scale tester.

If any one of the above items is met, it shall be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with psoriasis and healthy people
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | week0、week8、week16、week24
  PSQI is a 19-item self-rated questionnaire for evaluating subjective sleep quality over the previous month. A score above 5 suggests poor sleep quality.

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | week0、week8、week16、week24
  The PASI score ranges from 0 to 72, and the higher the score, the more serious the patient's condition. Generally speaking, a PASI score of less than 10 indicates mild psoriasis, 10-20 indicates moderate psoriasis, and more than 20 indicates severe psoriasis.
Dermatology Life Quality Index (DLQI) | week0、week8、week16、week24
  DLQI was a participant-reported questionnaire used to measure the health-related quality of life (QOL) of adults suffering from a skin disease. Scores ranged from 0-30, a higher score indicating a greater impact on a participant's QOL.
Visual Analogue Scale (VAS) | week0、week8、week16、week24
  The scoring criteria for pruritus level are as follows: absence of pruritus = 0; mild (intermittent itching, no scratching, no interference with daily activities) = 1-3 points; moderate (frequent itching, occasional scratching, impacting daily routine and sleep) = 4-6 points, and severe (intense itching, persistent scratching, significantly affecting daily life and sleep) = 7-10 points.
Hospital Anxiety and Depression Scale(HADS） | week0、week8、week16、week24
  For describing depression and anxiety in hospital patients

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality, China